CLINICAL TRIAL: NCT05352490
Title: Diagnosis of Heart Failure in Chronic Obstructive Pulmonary Disease Using the Lung Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: Lung ultrasound, COPD, HF
Record Dates: First submitted 2022-03-09; First posted 2022-04-28 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Dyspnea; Decompensated Heart Failure ; COPD Exacerbation
Keywords: COPD Acute Heart Failure Lung ultrasound
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF-group: patients with AECOPD and acute heart failure
  Interventions: Diagnostic Test: calculate LUS score
- non HF-group: patients with AECOPD without acute heart failure
  Interventions: Diagnostic Test: calculate LUS score

INTERVENTIONS:
Diagnostic Test: calculate LUS score — calculate LUS score

SUMMARY:
Acute Heart failure (AHF) is a common cause of acute exacerbation of chronic obstructive pulmonary disease (AECOPD). This association is frequently underestimated with regard to the difficulty of clinical diagnosis. The investigators expect that the application of the lung ultrasound could be useful in this issue.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a frequent disease in our population affecting mainly the elderly and males. Dyspnea is the most common reason for consultation for patients with COPD in ED. Distinguishing between pulmonary and/or cardiac origin can be challenging.Physical examination, laboratory findings and radiography are imperfect. Lung ultrasound sonography (LUS) has recently gained a large place in the diagnosis of heart failure (HF), but its contribution to the diagnosis of HF in COPD remains poorly studied.

Purpose: The purpose of this study is to assess the contribution of LUS in the diagnosis of HF in COPD patients with acute dyspnea

. Physical examination, laboratory findings and radiography are imperfect, resulting in a need for sophisticated test results that delay management. Lung ultrasonography is becoming a standard tool in critical cases in the ED. the investigators aim to perform ultrasonography on COPD patients admitted to the ICU with dyspnea, comparing lung ultrasonography results on initial presentation with the final diagnosis by the ICU team. Three items were assessed: artifacts (horizontal A lines or vertical B lines indicating interstitial syndrome), lung sliding, and alveolar consolidation and/or pleural effusion, these items were grouped to assess ultrasound profiles. This study assesses the potential of lung ultrasonography to diagnose heart failure.The second aim of this study was to evaluate the inter-observer reproducibility of LUS performed by ED residents in the evaluation of cardiac causes of acute dyspnea.This study includes patients with COPD consulting for acute dyspnea. We performed a lung ultrasound on all patients included. The diagnosis of heart failure (HF) was based on clinical, radiological, cardiac-ultrasound and expert data. The LUS diagnostic performance indicators were calculated using the different cut-off proposed by the LUS score.Then the probability of AHF was defined as : low probability (LUS<15) intermediate probability (15≤ LUS<30), and high probability (LUS≥30 ).

ELIGIBILITY:
Inclusion Criteria:

* patients with history of COPD admitted to the emergency department for dyspnea non traumatic dyspnea

Exclusion Criteria:

* instable hemodynamic or neurological status non consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with history of COPD admitted to the emergency departmet for dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
LUS in COPD patients whith pulmonory echography | 1day
  LUS measured whith pulmonory echography by the number of lines A and B.
the accuracy of LUS in the diagnosis of heart failure in COPD patients | 1day
  the accuracy of LUS in the diagnosis of heart failure in patients with COPD measured by area under the roc curve

CONTACTS AND LOCATIONS:
Overall Officials: Nouira semir Nouira semir, professor, Study Director — Principal Investigator university
Locations (1):
- Emergency Departement, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: official department website — http://www.urgencemonastir.com